CLINICAL TRIAL: NCT00431639
Title: The Effect of Animal-Assisted Therapy on Distress in Oncology Patients Being Treated for Pain
Brief Title: Effects of Pet Therapy on Pain in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 050093; 05-CC-0093; NCT00103688 (obsolete NCT alias)
Record Dates: First submitted 2007-02-03; First posted 2007-02-06 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2018-12-21

CONDITIONS: Cancer
Keywords: Animal-Assisted Therapy; Pain; Oncology; Cancer Pain
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Animal Assisted Therapy

ARMS (2):
- Comparison (Active Comparator): For the comparison condition, subjects will be asked to choose one of four topics that will be determined thatday with a recreational therapist for 20 minutes.
  Interventions: Behavioral: Animal Assisted Therapy
- Treatment (Active Comparator): The treatment condition will consist of a 20-minute visit by a therapy dog and its owner. Therapy dogowners will be instructed to limit conversation with the patient to topics of the therapy dog, thepatients pets, and pets in general.
  Interventions: Behavioral: Animal Assisted Therapy

INTERVENTIONS:
Behavioral: Animal Assisted Therapy — Every subject will be exposed to both treatment and comparison conditions.

SUMMARY:
This study will examine how animal-assisted therapy (AAT) affects aspects of pain. It will explore the possible benefits of the National Institutes of Health's AAT program on distress in cancer patients receiving pain and palliative care at the NIH Clinical Center. A number of studies on the benefits of patients interacting with companion animals have shown a positive effect of both pet ownership and AAT for patients with chronic illness. However, few such experimental studies have been conducted with cancer patients.

Patients 18 years of age and older who have been diagnosed with cancer and have been referred for consult with NIH's pain and palliative care team and recreation therapy may be eligible for this study.

Participants have two study sessions, each lasting about 20 minutes on two different days. In one session, they visit with an animal assistant therapy dog and its handler. In the other session they engage in a conversation that the patient identifies as non-stressful. Patients are asked to fill out four forms before and after each session with questions and statements about their pain, attitude towards pets, symptoms they might be having, and demographic information, such as age, sex, marital status, and so forth. On four separate occasions, 1 teaspoon of blood is drawn and a swab of saliva is collected from the mouth up to an hour after the session.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of the NIH Animal-Assisted Therapy (AAT) program on distress in oncology patients treated for pain. More than simply a physiologic or sensory response, pain is multidimensional. Pain management programs are best developed by selecting interventions based on the individual's pain experience. Strategies with several courses of action that complement each other may be selected to work together in a synergistic response to maximize pain relief. The goal of palliative care is to achieve the highest possible quality of life for patients, and indirectly, their families, through symptom control and attention to the whole patient: addressing physical, psychosocial, and emotional dimensions.

Limited research with persons receiving palliative care for cancer indicates that a variety of complementary interventions can mitigate psychological distress and improve quality of life (Ernst, 2001). A growing body of literature documenting positive effects of pet ownership and animal-assisted therapy (AAT) on patients with chronic illnesses warrants consideration of this type of intervention among the complementary approaches that may benefit terminally ill cancer patients.

The purpose of the proposed preliminary study is to explore the possible benefits of the existing NIH AAT program on psychological and physiological distress in cancer patients referred for pain and palliative care consults at the NIH Clinical Center. The primary outcome variable of interest is distress. Secondary outcomes of interest are pain intensity, pain unpleasantness, and use of pain medications. Attitudes towards pets is considered a moderating variable and will also be assessed.

A pre-post, within-subjects design will be used. Patients will be assigned in randomized block order to a comparison and treatment condition, administered at the same time of day on two consecutive days. The treatment condition is 20 minutes of AAT and the comparison condition is a 20-minute neutral discussion with a Recreational Therapist. All participants will be adult oncology patients consulted to the pain and palliative care service, and recreation therapy.

Psychological data will be collected pre and post session by survey instruments; medication use will be collected every 24 hours; physiological stress will be measured by salivary cortisol and, for patients with established indwelling catheters only, serum beta-endorphin levels.

Repeated measures ANOVA will be used to assess the effect of the two conditions (treatment vs. comparison) on each of the dependent variables. Descriptive statistics will be used to summarize baseline demographics.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

All adult cancer patients enrolled in research protocols who have a pain and palliative care consult, or a recreation therapy consult at the NIH Clinical Center may be eligible for the current study. Since the AAT provided at the NIH Clinical Center is generally available to the heterogeneous cancer population (with the exception of neutropenic patients) and the primary outcome of interest is distress regardless of the type of cancer, a heterogenous sample of cancer patients is considered appropriate for this investigation. While adults are the target population for this pilot study, if results are encouraging, minors will be considered for inclusion in subsequent studies.

INCLUSION CRITERIA:

* Ability to speak English and read at a 5th grade level
* 18 years of age or older
* Able to give informed consent
* Consulted to pain and palliative care team and Recreation Therapy
* Diagnosis of cancer

Available to be at the CRC on two consecutive days in the morning hours.

EXCLUSION CRITERIA:

* Interruption of primary protocol
* Allergies to or fear of dogs
* Patient on strict contact, or respiratory isolation restrictions
* Neutropenic patients

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-02-04; Primary Completion 2009-01-22 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Animal Assisted therapy on oncology patients being treated for pain | 72 hours
  Psychological and physiological distress is the primary outcome of interest in this study. This variable will be measured by two self report instruments, the Edmonton Symptom Assessment Scale and the Fear Visual Analog Scale, and two physiological assessments, salivary cortisol and serum beta endorphin. Several biochemical assays have been used as surrogate markers for stress. In this study, we propose to investigate two of these assays, serum beta-endorphin and salivary cortisol, in conjunction with other tools to assess levels of stress prior to, during and subsequent to treatment with animal-assisted therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Cohen Berger, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Friedmann E, Thomas SA. Pet ownership, social support, and one-year survival after acute myocardial infarction in the Cardiac Arrhythmia Suppression Trial (CAST). Am J Cardiol. 1995 Dec 15;76(17):1213-7. doi: 10.1016/s0002-9149(99)80343-9. PMID 7502998
- [Background] Barker SB, Pandurangi AK, Best AM. Effects of animal-assisted therapy on patients' anxiety, fear, and depression before ECT. J ECT. 2003 Mar;19(1):38-44. doi: 10.1097/00124509-200303000-00008. PMID 12621276